CLINICAL TRIAL: NCT04717440
Title: Assessment of the Reasons for Accepting or Refusing Early Palliative Care by the Patients Included in an Early Phase Clinical Trial
Brief Title: Assessment of the Reasons for Accepting or Refusing Early Palliative Care
Acronym: PALPHA-1
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET20-101 PALPHA-1
Record Dates: First submitted 2020-12-10; First posted 2021-01-22 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Cancer
Keywords: Cancer; Palliative care; Early phase trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients accepting palliative care: Patients included in an early phase trial and accepting palliative care
- Patients refusing palliative car: Patients included in an early phase trial but refusing palliative care

SUMMARY:
This is a prospective, multicentre study, considered as " non-RIPH ("Recherche n'Impliquant pas la Personne Humaine - Research that does not involve humans ". Indeed, the patient's participation in the study and the completion of the various questionnaires has no impact on patient's safety and is not likely to change patients' management. Patients accepting to take part to an early phase trial will be proposed to participate in the PALPHA-1 trial. They can accept or refuse to have palliative supportive care.

The main objective of this study is to assess the reasons for accepting and refusing early palliative care in patients included in an early phase clinical trial. The secondary objectives will enable to describe and analyze the number (effective) and the rate (%) of acceptance and/or refusal of early palliative support, to assess patients' understanding and perception of the " combined " management by comparing the semantic content of the patient-investigator ecological interaction during the proposal for inclusion in the trial (i.e. what was explicitly said), with that of the semi-structured post-consultation inclusion interviews ( ie what the patients understood, perceived), to compare the quality of life and the anxiety-depression of patients according to their acceptance or refusal of the mixed care at the inclusion and at the end of the early phase trial, to compare the clinical, medical and socio-demographic characteristics of the patients, the overall survival of patients according to their acceptance or refusal of the combined management and finally for the patients accepting the Palliative Care Management (PCM), to describe throughout the study, the patients' compliance to palliative supportive care undertaken.

DETAILED DESCRIPTION:
In a context of promotion of precision medicine, if palliative management and inclusion in an Early Clinical trial Phase (ECP) may at first glance appear antagonistic, some authors support the idea of a possible synergy in order to improve quality of life, reduce symptoms of exhaustion linked to treatment side effects and allow patients to complete their treatment protocol. To date and to our knowledge, few studies have assessed the brakes and/or levers for patient acceptance and/or refusal as well as the feasibility of a such mixed therapeutic management therapeutic. In this context, the beliefs and representations of patients must be taken into account in the decision-making process, which is also governed by the social norms of the caregiver-patient relationship. A better understanding of patients' acceptance and/or refusal of palliative care is an essential and innovative prerequisite for better understanding the processes involved at this stage of the care process.

The main objective of this study is to assess the reasons for accepting and refusing early palliative care in patients included in an early phase clinical trial. The secondary objectives will enable to describe and analyze the number (effective) and the rate (%) of acceptance and/or refusal of early palliative support, to assess patients' understanding and perception of the " mixed " management by comparing the semantic content of the patient-investigator ecological interaction during the proposal for inclusion in the trial (i.e. what was explicitly said), with that of the semi-structured post-consultation inclusion interviews ( ie what the patients understood, perceived), to compare the quality of life and the anxiety-depression of patients according to their acceptance or refusal of the mixed care at the inclusion and at the end of the early phase trial, to compare the clinical, medical and socio-demographic characteristics of the patients, the overall survival of patients according to their acceptance or refusal of the combined management and finally for the patients accepting the PCM, to describe throughout the study, the patients' compliance to palliative supportive care undertaken.

All patients approached for inclusion in an early phase clinical trial during the Multidisciplinary Consultation Meeting (MCR) will be offered to participate to the study. In order to assess the reasons for accepting / refusing the inclusion in palliative supportive care in patients entering an early phase clinical trial, two subgroups will be formed. The first group will be made up of patients who accepts joint palliative care (n = 20) and the second group of those who refuse (n = 20). Following their acceptance, the consultation for setting up the early phase clinical trial will be recorded and participants will be invited to participate in a semi-structured interview just before the first line of treatment. Patients (both having accepted or refused the palliative care) will also have to answer a self-questionnaire on quality of life and anxiety-depression at inclusion and at the end of the clinical trial. The study results will make it possible to determine patients' motivations for accepting or refusing palliative care management in order to better define their expectations, beliefs in terms of management, their understanding and impact of this management.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patient included in an early phase clinical trial
* Patient who has not been taken in charge for palliative care
* Life expectancy of at least 16 weeks
* Patient not opposed to data's collection and processing for the study
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient unable to read/understand the French language
* Patient with psychological disability (e.g. too great vulnerability, psychiatric disorder) or physical disability (e.g. physical / motor disability)
* Patients under autorship, curators or legal protection,
* Patients already participating in a clinical trial or interventional study related to supportive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multicentre study, considered as " non-RIPH (Recherche n'Impliquant pas la Personne Humaine - Research that does not involve humans ". Indeed, the patient's participation in the study and the completion of the various questionnaires has no impact on patient's safety and is not likely to change patient's management. Patients accepting to take part to an early phase trial will be proposed to participate in the PALPHA-1 trial. They can accept or refuse to have palliative supportive care. Patients' follow up will be performed according to the palliative standard procedures.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Assessment of the reasons for accepting / refusing early palliative care in patients included in an early phase clinical trial | At baseline
  Thematic content analysis of semi-directive qualitative interviews

SECONDARY OUTCOMES:
Description and analysis of the number (effective) of acceptance of early palliative support | At baseline
  Numbers of acceptance of the early palliative care management for all patients seen in early phase unit consultation
Description and analysis of the percentage of acceptance of early palliative support | At baseline
  Percentages of acceptance of the early palliative care management for all patients seen in early phase unit consultation
Assessment of patients' understanding and perception of the early palliative care management | At baseline
  Comparison of qualitative semantic content of patient-investigator interaction with the semi-directive post-consultation inclusion interview
Comparison of the quality of life of patients according to their acceptance or refusal of the mixed care | Up to 24 months
  Quality of life evaluated with the FACT-G7 (Functional Assessment of Cancer Therapy - General - 7-item version) questionnaire (range from 0 (better outcome) to 28 (worse outcome)
Comparison of the anxiety-depression of patients according to their acceptance or refusal of the mixed care | Up to 24 months
  Anxiety-depression evaluated with the HADS (Hospital Anxiety and Depression Scale) questionnaire (range 0-7: No symptoms, range 8-10: Doubtful symptoms, range >=11: Symptoms of anxiety or depression)
Comparison of the clinical, medical and socio-demographic characteristics of patients for the patients accepting the palliative care management | At baseline
  Using PALLIA 10 scale (PALLIAtive scale composed of 10 items, minimum value: 1, maximum value: 10. A specialized advice in palliative care is required if score > 3)
Comparison of the clinical, medical and socio-demographic characteristics of patients who accept or refuse the palliative care management | At baseline
  Using PRONOPALL score (Prognostic overall survival score). Range 0-3: Favorable overall survival score, Range 4-7: Intermediate overall survival score, Range 8-10: Unfavorable overall survival score.
Comparison of the clinical characteristics of patients who accept or refuse the palliative care management | At baseline
  Clinical symptoms evaluated using ESAS (Edmonton Symptom Assessment System) questionnaire (range from 0 (better outcome) to 10 (worse outcome))
Comparison of the socio-demographic characteristics of patients who accept or refuse the palliative care management | At baseline
  Patients' characteristics (Age, sex, family situation, place of residence, socio-educational level, professional activity)
Comparison of the medical characteristics of patients who accept or refuse the palliative care management | Up to 24 months
  Patients' medical history: Treatments
Comparison of the medical characteristics of patients who accept or refuse the palliative care management | Up to 24 months
  Patients' medical history: Use of specialists' consultations (e.g. intensive care unit, emergency hospitalization, palliative care unit, number/types of consultations, pain, nutrition)
Comparison of the use of social services of patients who accept or refuse the palliative care management | Up to 24 months
  Patients' medical history: Use of social service...
Overall survival of patients according to their acceptance or refusal of the "mixed" management | Up to 24 months
  Vital status
For patients having accepted the palliative support, description throughout the study of patients' compliance to palliative supportive care undertaken | Up to 24 months
  Patients having performed at least 50 percent of the visits

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle CHVETZOFF, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Derived] Chvetzoff G, Girodet M, Despax J, Baudry V, Duranti J, Mastroianni B, Vanacker H, Vinceneux A, Brahmi M, Renard O, Gautier J, Britel M, Ducimetiere F, Anota A, Cassier P, Christophe V. Reasons for acceptance and refusal of early palliative care in patients included in early-phase clinical trials in a regional comprehensive cancer centre in France: protocol for a qualitative study. BMJ Open. 2022 Apr 22;12(4):e060317. doi: 10.1136/bmjopen-2021-060317. PMID 35459679